CLINICAL TRIAL: NCT04000425
Title: Evaluating Potential Clinical Utilities of Circulating Tumor DNA in Gastric Cancer
Brief Title: Potential Clinical Utilities of Circulating Tumor DNA in Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZSGC-005
Record Dates: First submitted 2019-06-26; First posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Circulating Tumor DNA; Minimal Residue Disease; Chemotherapy Response
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ctDNA detection: The blood samples for ctDNA and other tumor markers (such as CEA, et al.) will be first collected within 7 days before surgery, and then be tested after radical gastrectomy in scheduled interval.
  Interventions: Combination Product: AVENIO ctDNA surveillance kit

INTERVENTIONS:
Combination Product: AVENIO ctDNA surveillance kit — AVENIO circulating tumor DNA (ctDNA) Analysis Kits is a portfolio of three next-generation sequencing (NGS) liquid biopsy assay kits for oncology research: the AVENIO ctDNA Targeted Kit, Expanded Kit and Surveillance Kit.

SUMMARY:
This study is designed to evaluate the potential clinical utility of ctDNA in the field of gastric cancer treatment,especially the usage of an indicator of MRD(minimal residual disease) in post radical gastrectomy patients. The primary purpose of this trial is to demonstrate if the postoperative ctDNA analysis could be used as an indicator of MRD or adjuvant chemotherapy response in advanced gastric cancer after radical gastrectomy.The second purpose is to describe the profile of ctDNA in gastric cancer.

DETAILED DESCRIPTION:
Gastric cancer is an important health problem, being the fifth most common cancer and the third leading cause of cancer related death worldwide.Incidence shows clear regional and sex variations-rates are highest in Eastern Asia, Eastern Europe, and South America and lowest in Northern and Southern Africa. In China, gastric cancer accounts for nearly 16% of all malignant tumors and more than 80% of gastric cancer are in advanced stage.

Minimal residual disease (MRD) was proposed to describe the remaining tumor cells after treatment with curative intent. For curable gastric cancer, MRD means residential cancer cells after radical gastrectomy which share phenotypic similarity and genetic heritage with the original tumor. Treating MRD can increase the rates of cure had been supported by the experience of using adjuvant therapy for some type of solid tumor (for example, colorectal cancer, breast cancer). The challenge in monitoring the MRD in gastric cancer patients is that there is no very sensitive method. Computed tomography(CT) and blood tumor markers are either difficult to detect peritonial dissemination, the most frequent recurrent pattern in gastric caner or with limited sensitivity and specificity.

Tumor-specific DNA mutations detected in the cell-free component of peripheral blood, which is known as circulating tumor DNA (ctDNA), in most patients, allow for the noninvasive molecular characterization detection of tumors, including genetic changes that are revealed by the selective pressure of adjuvant therapies. Considering the origin of ctDNA, it can be from different subclones of primary tumor or both primary and metastatic tumors, the ctDNA may overcome the problems caused by tumor heterogeneity. Additionally, the short half-life of ctDNA, about 2 hours, makes ctDNA an ideal dynamic marker of tumor bulk.

In summary, the ctDNA is a good candidate to be a new kind of blood tumor marker. The preliminary studies had shown very good prospects in some tumors, including breast caner and colon cancer.But little was known in gastric cancer, so we designed this study to demonstrate the potential clinical utility of ctDNA in the field of gastric cancer treatment, especially the usage of an indicator of MRD in post radical gastrectomy patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients age 18 - 75.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0,1 or 2.
3. Histologically proven primary stomach adenocarcinoma with Lauren type by gastroscopic biopsy before operation.
4. Clinical stage is cT3/4N+M0 and the tumor is resectable in initial evaluation.
5. No preoperative tumor therapy, including chemotherapy, radiotherapy, et al.
6. No concomitant other malignant tumor or treated malignant tumor within last five years.
7. Signed informed consent.
8. Consent to provide research blood/tissue samples and clinicopathological information.

Exclusion Criteria:

1. Radical gastrectomy was found cannot be achieved during operation due to metastasis or adjacent organ invasion.
2. Only preoperative or postoperative blood sample was harvest or qualified.
3. No qualified paired tissue samples.
4. No complete clinicopatholoical information and follow-up.
5. Presence of any systemic illness incompatible with participation in the clinical trial or inability to provide written informed consent.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Stomach adenocarcinoma patients who plan to receive radical gastrectomy and continuous circulating tumor DNA monitoring
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Description of disease recurrence risk according to first positive ctDNA detection | 2 years
  Time is measured from first positive ctDNA detection to disease-free survival event.
Description of ctDNA changing to adjuvant chemotherapy response | 2 years
  For subjects with postoperative positive ctDNA, time is measured from first adjuvant chemotherapy to first negative ctDNA detection.

SECONDARY OUTCOMES:
Leading time between ctDNA detection and disease recurrence detected by conventional methods | 2 years
  Time is measured between first positive ctDNA detection and first recurrence detected by conventional methods.
The ctDNA level/mutations in gastric cancer preoperatively | Within 7 days before operation
  Profiling of the most frequently detected gene mutations and level of mutations in preoperative ctDNA.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoqing Tang, MD, Principal Investigator — Fudan University
Locations (1):
- ZhongShan hospital FuDan university, Shanghai, Shanghai Municipality, China